CLINICAL TRIAL: NCT04618042
Title: FX06 to Rescue Acute Respiratory Distress Syndrome During Covid-19 Pneumonia
Acronym: FX-COVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP200495; 2020-002056-20 (EudraCT Number)
Record Dates: First submitted 2020-10-23; First posted 2020-11-05 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Ards; Covid19; Pneumonia
Keywords: FX06; Pulmonary vascular hyperpermeability
MeSH Terms: conditions — Acute Lung Injury; COVID-19; Pneumonia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FX06 (Experimental)
  Interventions: Drug: FX06
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo of FX06

INTERVENTIONS:
Drug: FX06 — FX06 i.v.: 400 mg per day (divided in two injections) during 5 days
  Arms: FX06
Drug: Placebo of FX06 — Placebo i.v.: 400 mg per day (divided in two injections) during 5 days
  Arms: Placebo

SUMMARY:
Vascular leakage following endothelial injury, responsible for interstitial and alveolar edema, is a major feature of pathogen induced acute lung injury. As acute respiratory distress syndrome (ARDS) due to pandemic Covid-19 is associated with more than 60% mortality, controlling vascular leakage may be a major target to decrease the mortality associated with the spreading of the disease in France.

FX06, a drug under clinical development containing fibrin-derived peptide beta15-42, is able to stabilize cell-cell interactions, thereby reducing vascular leak and mortality in several animal models, particularly during lipopolysaccharide-induced and dengue hemorrhagic shock . A phase I study was conducted in humans, with no specific adverse event detected with a dose up to 17.5 mg/kg. In a phase II randomized multicentre double-blinded trial in 234 patients suffering from ST+ acute coronary syndrome, FX06 treated patients exhibited a 58% decrease in the early necrotic core zone. Importantly, adverse events were highly comparable between groups, indicating a high safety profile for the drug . Lastly, the drug was used as a salvage therapy in a patient exhibiting a severe ARDS following EBOLA virus infection . Altogether, those data indicate that FX06 is well tolerated in humans and is a potent regulator of vascular leakage.

Our hypothesis here is that FX06 may decrease pulmonary vascular hyperpermeability during ARDS following SARS-CoV-2 infection, thereby improving gas exchanges and the outcome of infected patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. SARS-CoV-2 induced pneumonia confirmed by a positive PCR test in nasopharyngeal swab or respiratory tract secretions and ≤ 85 years
3. Acute respiratory distress syndrome (ARDS) according to Berlin criteria (bilateral pulmonary infiltrates on frontal chest x-ray, PaO2/FiO2 ratio ≤300 mmHg, objective assessment excluding hydrostatic pulmonary edema)
4. Need for endotracheal intubation and mechanical ventilation
5. Informed consent by patient or legal representative. According to the specifications of emergency consent, randomization without the close relative or surrogate consent could be performed.
6. Affiliated to a social security system
7. Highly effective method of contraception and negative highly sensitive pregnancy test, for women of childbearing potential

Exclusion Criteria:

1. Mechanically ventilation for more than 4 days
2. Patient receiving drugs interfering with inflammation: Non-steroidal anti-inflammatory drugs, immunoglobulins.
3. Patients receiving chemotherapy, radiotherapy or immunotherapy for malignancy
4. Participation in another interventional clinical trial
5. Pregnant or lactating women
6. Patient moribund on the day of randomization, defined by a SAPS-II score>90
7. Contra-indication for vascular access implantation for transpulmonary thermodilution monitoring
8. Severe or terminal renal insufficiency (creatinine clearance <30 ml/min)
9. Severe hepatic insufficiency (hepatic SOFA score>2)
10. Severe cardiac insufficiency, with left ventricular ejection fraction<30%
11. Any history of severe allergic drug reaction (anaphylactic shock or allergic angioedema)
12. Persons deprived of their liberty by a judicial or administrative decision (guardianship or tutelage measure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-06-13 (Actual)

PRIMARY OUTCOMES:
Change in extravascular lung water index (EVLWi) | Between Day 1 and Day 7
  Assessed by transpulmonary thermodilution Transpulmonary thermodilution systems, part of the standard management in ICU, allow a direct evaluation of vascular hyperpermeability in the lungs using thermodilution technique. EVLWi is a reliable parameter, independently associated with mortality during ARDS

SECONDARY OUTCOMES:
Evolution of daily extravascular lung water index (EVLWi) | Between Day 1 and Day 7
  measured by transpulmonary thermodilution during 7 days
Evolution of daily cardiac index | Between Day 1 and Day 7
  measured by transpulmonary thermodilution during 7 days
Evolution of global end-diastolic volume index | Between Day 1 and Day 7
  measured by transpulmonary thermodilution during 7 days
Evolution of pulmonary vascular permeability index | Between Day 1 and Day 7
  measured by transpulmonary thermodilution during 7 days
Overall survival | Day 30
Mortality rate in ICU and in hospital | Through study completion an average of 2 months
Rate of withdraw or withhold life-sustaining treatments decision | Day 30
Daily weight | Between Day 1 and Day 7
Daily fluid balance | Between Day 1 and Day 7
Evolution of albuminemia | Between Day 1 and Day 7
  Evolution of blood biological criteria (g/L)
Duration of mechanical ventilation | Day 30
Proportion of participants alive and off invasive mechanical ventilation | Day 30
Evolution of Murray ARDS severity score | Day 1 to day 15
Evolution of radiological Weinberg score | Day 1 to Day 30
  Scale from 0 to 12 better with higher score indicating more severe radiological pulmonary severity
Evolution of pulmonary Sequential Organ Failure Assessment) score. | Day 1 to day 15
  Scale from 0 to 4 betterwith higher score indicating more severe pulmonary disease
Rate of rescue therapy with Veino-veinous V-ECMO | Through study completion an average of 2 months
Evolution of SOFA (Sequential Organ Failure Assessment) score | Day 15
  Scale from 0 to 24, lower is better.
Organ failure free days | Day 15
  one or more SOFA sub-score >=3
Renal replacement therapy free days | Day 30
Duration of renal replacement therapy free days | Day 30
Nature and frequency of adverse events | Through study completion an average of 2 months
Evolution of FX06 concentration | Day 1
  measured at day 1 at time 0 (before FX06 application) and after 5, 15, 30, 60 min
Immunogenicity (antibody against FX06) induced by the drug, performed by ELISA according to manufacturer's procedure | Day 7
  A test for immunogenicity will be performed on a serum sample at day 7 (2 days after the end of treatment administration) to detect any antibody against FX06. The assay will consist in a three-fold procedure, as recommended by the manufacturer. An initial screening assay will qualitatively measure antibodies to FX06. Samples deemed positive will be subject to a confirmatory assay, which will determine the specificity of the detected antibody against FX06. The third tier of the assay will consist in titre analysis to semi-quantitatively assess the antibody response.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Service de Médecine Intensive Réanimation - CHU Angers, Angers
  - Service de Médecine Intensive Réanimation - CHI de Poissy, Chambourcy
  - Hôpital Pitié Salpêtrière, Paris

REFERENCES:
- [Derived] Guerin E, Belin L, Franchineau G, Le Guennec L, Hajage D, Diallo MH, Frapard T, Le Fevre L, Luyt CE, Combes A, Germain S, Hayon J, Asfar P, Brechot N. FX06 to rescue SARS-CoV-2-induced acute respiratory distress syndrome: a randomized clinical trial. Crit Care. 2023 Aug 29;27(1):331. doi: 10.1186/s13054-023-04616-1. PMID 37641136